CLINICAL TRIAL: NCT00447642
Title: A Multi-center, Placebo-Controlled, Randomized, Parallel-Group, Dose-Ranging Study to Assess the Efficacy and Safety of LX201 Implantation for the Prevention of Corneal Allograft Rejection Episodes or Graft Failure in Subjects Who Have Experienced One or More Rejection Episodes Following Penetrating Keratoplasty
Brief Title: Study to Assess LX201 for Prevention of Corneal Allograft Rejection or Graft Failure in Subjects Who Have Experienced One or More Rejection Episodes Following Penetrating Keratoplasty
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The primary efficacy endpoint was not met
Sponsor: Lux Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LX201-02
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Corneal Transplantation; Corneal Graft Rejection
Keywords: immunology; cornea; allograft; corneal allograft rejection; graft failure
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LX201 0.50 inch implant (Experimental): LX201 implant contained 30% cyclosporine A by weight and 0.50 inch in length
  Interventions: Drug: LX201
- LX201 0.75 inch implant (Experimental): LX201 implant contained 30% cyclosporine A by weight and 0.75 inch by length
  Interventions: Drug: LX201
- Placebo 0.75 inch implant (Placebo Comparator): Silicone implant not containing cyclosporine A, 0.75 inch in length
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LX201 — LX201 was a novel sustained-release silicone implant containing 30% cyclosporine A by weight.
  LX201 was available in two different lengths, 0.50 and 0.75 inch. Each implant is 0.08 inch wide and 0.04 inch in height. The implants are flat on one side (the posterior surface, which is applied to the episclera) and the anterior surface and ends were rounded.
  Arms: LX201 0.50 inch implant; LX201 0.75 inch implant
Other: Placebo — The placebo was a silicone implant 0.75 inch in length. It contained no cyclosporine A
  Arms: Placebo 0.75 inch implant

SUMMARY:
This study will evaluate the use of LX201 to prevent future graft rejection episodes and/or graft failure in patients who have undergone corneal transplantation and who have recently experienced a rejection episode due to an immune response.

DETAILED DESCRIPTION:
LX201 was a novel sustained-release silicone implant containing 30% cyclosporine A by weight. LX201 is intended for surgical episcleral placement in the eye.

The study was a Phase 2/3, multi-center, placebo-controlled, randomized, parallel-group, dose-ranging study of LX201 for prevention of corneal allograft rejection or graft failure in subjects who have had one or more rejection episodes following penetrating keratoplasty.

After Visit 12 (Week 52), subjects in the USA and India with the implant in the study eye were to be followed for safety at least once per year for a 2 year period or until time of implant removal. In Germany, the implant was to be removed at Week 52 with a 3-month safety follow-up period after removal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, within 6 months prior to study randomization, have experienced 1 or more corneal allograft rejection episodes following penetrating keratoplasty
* Must be on a stable medical regimen for at least 14 days at the time of randomization into the study
* Conjunctiva must be suitable for implantation with the study device

Exclusion Criteria:

* Any condition that would greatly increase the risk of non-rejection graft failure such as Stevens-Johnson syndrome, xerophthalmia or severe exposure keratitis.
* Schirmer's test ≤ 5 mm in 1 minute.
* Clinical evidence of limbal stem cell deficiency.
* History of or active herpes simplex virus keratitis or other acute corneal infection
* Subjects who have had > 3 failed grafts in the ipsilateral eye
* Uncontrolled glaucoma as evidenced by an intraocular pressure of > 21 mmHg while on maximal medical therapy
* Clinically suspected or confirmed ocular lymphoma
* Treatment with a systemic immunosuppressive regimen within the previous 30 days; systemic prednisone (or its equivalent) of ≤ 10 mg daily is, however, permitted.
* Any implantable corticosteroid-eluting device (e.g., Retisert™, Posurdex®, Medidur™, I-vation™ triamcinolone acetonide [TA] intravitreal implant)
* Subjects who periodically require high-dose systemic steroid treatment (e.g., for exacerbation of chronic obstructive pulmonary disease).
* Subjects who have received treatment with a monoclonal antibody or any other biologic therapy within the previous 90 days or alemtuzumab within the previous 12 months
* History of herpes zoster or varicella infection within 6 weeks prior to enrollment, or chicken pox exposure within 21 days before enrollment
* Seropositivity for human immunodeficiency virus (HIV)
* Previous exposure or known contraindication to administration of cyclosporine
* Recipients of a solid organ transplant
* Currently participating in another clinical trial with an investigational agent in the 30 days prior to study participation and/or has not recovered from any reversible effects or side effects of prior investigational agent
* Currently pregnant or lactating
* Active, extraocular and/or systemic infection requiring the prolonged or chronic use of antimicrobial agents or the presence of active hepatitis A, B or C
* Current malignancy or a history of malignancy (within the previous 5 years) except non-metastatic basal or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix that has been treated successfully
* Active peptic ulcer disease
* Co-morbid conditions that require immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
prevention of corneal allograft rejection or graft failure | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Anglade, MD, Study Chair — Chief Medical Officer, Lux Biosciences, Inc.
Locations (30):
- United States (24):
  - Cornea Consultants of Arizona, Phoenix, Arizona
  - Loma Linda University Health Care, Loma Linda, California
  - USC Doheny Eye Institute, Los Angeles, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Emory Eye Center, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Price Vision Group, Indianapolis, Indiana
  - The Eye Center at Union Memorial Hospital, Baltimore, Maryland
  - Wilmer Eye Institute, Cornea Service, Baltimore, Maryland
  - New England Eye Center, Boston, Massachusetts
  - W.K. Kellogg Eye Center - University of Michigan, Ann Arbor, Michigan
  - MN Eye Consultants, P.A., Bloomington, Minnesota
  - Tauber Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - UMDNJ - New Jersey Medical School Institute of Ophthalmology and Visual Science, Newark, New Jersey
  - New York Eye and Ear Infirmary, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Cornea Consultants of Albany, Slingerlands, New York
  - Duke University Eye Center, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cornea Associates of Texas, Dallas, Texas
  - Virginia Eye Consultants, Norfolk, Virginia
  - Eye Associates NW, Seattle, Washington
- Germany (6):
  - Augenklinik, Universitat Erlangen-Nurnberg, Erlangen
  - Cornea Bank, Universitätsklinikum Essen, Essen
  - Klinik fuer Ophthalmologie Campus Kiel, Kiel
  - Ludwig Maximilians Universität, München
  - Augenklinik der Technischen Universität München, München
  - Augenklinik Wuerzburg, Würzburg